CLINICAL TRIAL: NCT00965016
Title: The Therapeutic Effect of Induced Hypothermia in Cardiac Arrest Patients Rescued by Extracorporeal Cardiopulmonary Resuscitation (ECPR).
Brief Title: Induced Hypothermia in Cardiac Arrest Patients Rescued by Extracorporeal Cardiopulmonary Resuscitation.
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Min-Sheng General Hospital (Other)
Responsible Party: Yao, Director of department of Education, Min-Sheng General Hospital
Allocation: Non-Randomized | Model: Factorial | Masking: None | Purpose: Treatment
Other Study IDs: MSEIRB0980106
Record Dates: First submitted 2009-08-23; First posted 2009-08-25 (Estimated); Last update posted 2009-08-25 (Estimated); Status verified 2009-08

CONDITIONS: Out-of-Hospital Cardiac Arrest
Keywords: Extracorporeal membrane oxygenation，induced hypothermia
MeSH Terms: conditions — Out-of-Hospital Cardiac Arrest

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- No Hypothermia, No intervention, ECMO (Sham Comparator): No hypothermia used during ECPR
  Interventions: Procedure: hypothermia
- Hypothermia, intervention, ECMO (Active Comparator): Hypothermia + intervention
  Interventions: Procedure: hypothermia
- Hypothermia, no intervention, ECMO (Active Comparator): Hypothermia without intervention after ECMO
  Interventions: Procedure: hypothermia

INTERVENTIONS:
Procedure: hypothermia — Core temperature --> 34.9℃ within 30 min --> 33.5℃ within 120min --> 33℃for 24 H Decrease temperature in 0.9℃/hour
  Other Names: ECPR

SUMMARY:
Background： Cardiopulmonary resuscitation (CPR) with closed-chest cardiac massage has been shown that survival to discharge rate is poor. Attempt to increase success, some aggressive methods such as extracorporeal membrane oxygenation (ECMO) has been used (also known as extracorporeal cardiopulmonary resuscitation, ECPR). Otherwise, anoxic brain injury is another issue after CPR. In recent years, some randomized prospective controlled trials of induced hypothermia (IH) to 33℃ for 12 to 24 hours has been demonstrated to significantly improve outcome in cardiac arrest patients. Because ECMO also could provide hypothermia management, we plan this study to evaluate the cerebroprotective effect of ECPR with induced hypothermia. We will try to analyze risk factors influencing patient survival and weaning from ECPR and the optimal management for this ominous prognosis group.

Method:

The patients were recruited into the ECPR group only if they:

1. in cardiac arrest that necessitated external or open-chest cardiac massage and a large amount of epinephrine (>5 mg) during CPR.
2. Could not be returned to spontaneous circulation within 10 to 20 min. After ECPR, the body temperature was started to be cooled down. Within 3 hours, the patients have been well studied to search for potential reason of CPR. If the patients have no heart problem or only intervention needed, they can be grouped into 1. Group 2 is the group, which some further operation must be delivered. Group 3 is the group who cannot afford to receive hypothermia (The physician in charge don't agree the trial.) In ECMO-supported patients, two resulting comparisons were of concern: 1) ECMO weaning versus nonweaning and 2) survival-to-discharge versus in-hospital death. We attempted to identify the risk factors that affected weaning and survival, and we analyzed the effect of ECPR with hypothermia on survival.

Expected result:

We will prove ECPR with hypothermia is a perfect strategy. And within three groups of the patients, ECMO +induced hypothermia will be the most optimal choice.

DETAILED DESCRIPTION:
Induced Hypothermia Protocol for comatose patient from CPR Core temperature: 34.9℃ within 30 min, 33.5℃ within 120min and 33℃ for 12-24 Hours

* Decrease temperature in 0.9℃/hour
* CVP monitoring
* the infusions were temporarily stopped if CVP increased > 5 mm Hg over 5 mins.
* Continuous temperature monitoring with a rectal probe or bladder catheter
* One must be vigilant to avoid k+, Ma2+, and P depletion during and immediately after the infusion, particularly given the increased risk of cardiac arrhythmia that occurs with induced hypothermia.
* An evaluation of neurologic status
* IV Dormicum (midazolam 2 to 5 mg或0.125 mg/kg/hr initially) and fentanyl (0.002 mg/kg/hr initially), Pavulon (pancuronium 0.1 mg/kg) every 2 hours for a total of 32 hours.
* ABG values were used to adjust the ventilator to maintain PaO2>100 mm Hg and PaCO2<40 mm Hg.
* MAP: 90 ~ 100 mm Hg
* Lidocaine bolus (1 mg/kg) followed by an infusion (2 mg/min for 24 hours)
* K+> 4.0 mmol/L
* RI infusion < 180 mg/deciliter (10 mmol per liter)
* Antibiotics with β-lactam；Aspirin
* The temperature was maintained at 33℃ for 24 hours from the start of cooling, followed by passive rewarming, which we expected would occur over a period of 8 hours, followed by active rewarming.

ELIGIBILITY:
Inclusion Criteria:

* 1. in cardiac arrest that necessitated external or open-chest cardiac massage and a large amount of epinephrine (>5 mg) during CPR.
* 2. Could not be returned to spontaneous circulation within 10 to 20 min

Exclusion Criteria:

* contraindicated to ECMO use

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 45 (Estimated)
Dates: Start 2009-01; Primary Completion 2009-12 (Estimated); Study Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
1) ECMO weaning versus nonweaning and 2) survival-to-discharge versus in-hospital death. | 20091231

SECONDARY OUTCOMES:
Brain injury | 20091231

CONTACTS AND LOCATIONS:
Overall Officials: Shaojung Li, physician, Principal Investigator — Director, department of cardiovascular surgery
Locations (1):
- Min-sheng General Hospital, Taoyuan District, Taiwan